CLINICAL TRIAL: NCT00638703
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Multi-center, International Study to Evaluate the Efficacy and Safety of OxabactTM to Reduce Urinary Oxalate in Subjects With Primary Hyperoxaluria
Brief Title: Study to Evaluate the Efficacy and Safety of OxabactTM on Reduction of Urinary Oxalate in Primary Hyperoxaluria Patients
Acronym: PHOENIX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: OxThera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC3-DB-01; DB-01
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2011-06

CONDITIONS: Primary Hyperoxaluria
Keywords: hyperoxaluria; PH; oxalate
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Size 2 enteric coated capsule containg lyophilized Oxalobacter formigenes
  Interventions: Biological: Oxalobacter formigenes
- II (Placebo Comparator): Size 2 enteric coated capsule containg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Oxalobacter formigenes — NLT (not less than) 10^7 CFU Oxalobacter formigenes twice daily for 24 weeks
  Other Names: - Oxabact(tm); - OC3
  Arms: I
Drug: Placebo — placebo
  Arms: II

SUMMARY:
The main purpose of this study is to determine if Oxalobacter formigenes is effective at lowering urinary oxalate levels in patients with primary hyperoxaluria.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (or legally acceptable representative) must give written informed consent (and assent for subjects ≥ 12 years or country specific age as appropriate). For subjects less than 18 years of age, parent or guardian will provide informed consent and the subject will provide witnessed verbal assent
2. Male or female subjects ≥ 5 years of age
3. Urinary oxalate excretion of > 1.0 mmol/1.73m2/day at Baseline
4. Documentation of diagnosis of PH I or PH II by any one of the following:

   1. Liver biopsy confirmation of deficient liver specific peroxisomal alanine-glyoxylate aminotransferase, (AGT) or mislocalization of AGT from peroxisomes to mitochondria (PH I) or deficient glyoxylate reductase/hydroxypyruvate reductase (GR/HPR) activity (PH II)
   2. Homozygosity or compound heterozygosity for a known mutation in the causative genes for PH I and PH II
   3. Increased glycolate excretion for PH I or increased L-glycerate excretion for PH II
5. Subjects receiving pyridoxine must be receiving a stable dose for at least 3 months prior to entry in to the study and must remain on the stable dose during the study. Other (non-pyridoxine naïve) subjects (e.g. Pyridoxine non-responder: <30% reduction of the urine oxalate levels) not receiving pyridoxine at study entry must be willing to refrain from initiating pyridoxine during study participation. Note: There will be no pyridoxine-naïve subjects enrolled in the study.
6. Renal function defined as an estimated GFR ≥ 50 ml/min normalized to 1.73m2 body surface area

Exclusion Criteria:

1. Pregnant, lactating, or actively menstruating women and women of child-bearing potential who are not using adequate contraceptive precautions. Sexually active females, unless surgically sterile or at least 2 years post-menopausal, must be using a highly effective contraception (including oral, transdermal, injectable, or implanted contraceptives, IUD, abstinence, use of a condom by the sexual partner, or sterile sexual partner) for 30 days prior to the first dose of OxabactTM and must agree to continue using such precautions during the clinical study.

   Note: A highly effective method of birth control is defined as one that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomised partner.
2. Positive serum pregnancy test.
3. Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to randomization or not willing to forego other forms of investigational treatment during this study.
4. Subjects on hemodialysis or peritoneal dialysis.
5. Subjects who have undergone transplantation (solid organ or bone marrow).
6. Chronic gastrointestinal disease associated with enteric hyperoxaluria, e.g. history of inflammatory bowel disease, colostomy. Note: For clarity, existence of Secondary Hyperoxaluria (e.g. with cystic fibrosis, chronic inflammatory bowel diseases, short bowel syndrome and/or deficiency of intestinal oxalate-degrading bacteria is included (as an exclusion criteria).
7. Current systemic (oral, IM, IV) antibiotic use or received systemic antibiotics within 14 days of study enrolment.
8. History of chronic, recurrent infections requiring >2 courses of antibiotics in the past 6 months.
9. History of malignancy except for basal or squamous cell skin cancer that has been excised.
10. Unable to collect 24-hour urine samples or follow other study procedures.
11. Subjects who cannot swallow a size 2 capsule.
12. Presence of a medical condition that the Principal Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures.
13. Subjects who require immune suppressive therapy (including prednisone of > 10mg daily for more than 2 weeks).
14. Subjects from correctional facilities or asylums.
15. Subjects who are mentally handicapped.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction in urinary oxalate Percentage change in urinary oxalate (expressed as mmole/1.73m2 /day) from Baseline to Week 24 | 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects who are responders at Week 24 where response is defined as a 20% or greater reduction from Baseline urinary oxalate to Week 24 | 24 weeks
Percentage change in urinary oxalate (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 | 24 weeks
Percentage change in urinary oxalate (expressed as mmole/1.73m2/day and as molar oxalate to creatinine ratio) from Baseline to Week 12 | 12 weeks
Percentage change in urinary oxalate (expressed as mmole/1.73m2/day and as molar oxalate to creatinine ratio) from Baseline to average of Weeks 12 and 24 | 12 and 24 weeks
Frequency of AEs and SAEs | over 24 weeks
Laborator safety data | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Milliner, M.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic (Department of Pediatric Nephrology), Rochester, Minnesota, United States